CLINICAL TRIAL: NCT00006360
Title: Conformal and Intensity Modulated Irradiation for Oropharyngeal Cancer
Brief Title: Radiation Therapy in Treating Patients With Stage II or Stage III Oropharyngeal Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: RTOG-0022; CDR0000068231; RTOG-H-0022
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2016-12

CONDITIONS: Head and Neck Cancer; Radiation Toxicity
Keywords: stage II squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; radiation toxicity
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries; Squamous Cell Carcinoma of Head and Neck | interventions — Radiation Protection; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: radioprotection
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiation therapy in treating patients who have stage II or stage III oropharyngeal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess target coverage and major salivary gland sparing in patients with stage II or III oropharyngeal cancer treated with intensity-modulated radiotherapy.
* Determine the nature and prevalence of acute and late side effects of this treatment in these patients.
* Determine the rate and pattern of locoregional tumor recurrence in these patients after this treatment.

OUTLINE: This is a multicenter study.

Patients receive 3-D conformal radiotherapy and/or intensity-modulated radiotherapy daily 5 days a week for 6 weeks, in an effort to spare major salivary glands.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 57-64 patients will be accrued for this study over 27 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage II or III (T1-T2, N0-N1) squamous cell carcinoma of the oropharynx (tonsil, base of tongue, or palate)

  * Lymph nodes in both sides of neck at risk of metastatic disease and require radiotherapy
  * Patients upstaged by imaging to N2 are eligible
* Measurable or evaluable disease

  * Greater than 1 cm in one dimension or with necrotic regions if by CT or MRI scan
* Surgery of the primary tumor or lymph nodes limited to incisional or excisional biopsies
* No distant metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* Zubrod 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No active untreated infection
* No other malignancy within the past 5 years except nonmelanoma skin cancer or a carcinoma not of head or neck origin
* No concurrent major medical or psychiatric illness that would preclude study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* More than 3 months since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior head or neck radiotherapy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent treatment for head and neck cancer
* No prophylactic amifostine or pilocarpine

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-02; Primary Completion 2005-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Acute salivary gland toxicity
Locoregional control
Whole mouth saliva output relative to pre-radiotherapy measurements
Acute mucositis and other acute and late toxicities

CONTACTS AND LOCATIONS:
Overall Officials: Avraham Eisbruch, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (18):
- United States (15):
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - Community Regional Cancer Center at Community Medical Center, Toms River, New Jersey
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - Community Cancer Center at Rutland Regional Medical Center, Rutland, Vermont
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
- Canada (3):
  - Stollery Children's Hospital at University of Alberta Hospital, Edmonton, Alberta
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Background] Ploquin N, Lau H, Dunscombe P. Intensity modulated and three-dimensional conformal radiation therapy plans for oropharyngeal cancer: a comparison of their sensitivity to set-up errors and uncertainties. Curr Oncol. 2006 Apr;13(2):61-6. doi: 10.3390/curroncol13020005. PMID 17576443
- [Result] Eisbruch A, Harris J, Garden AS, Chao CK, Straube W, Harari PM, Sanguineti G, Jones CU, Bosch WR, Ang KK. Multi-institutional trial of accelerated hypofractionated intensity-modulated radiation therapy for early-stage oropharyngeal cancer (RTOG 00-22). Int J Radiat Oncol Biol Phys. 2010 Apr;76(5):1333-8. doi: 10.1016/j.ijrobp.2009.04.011. Epub 2009 Jun 18. PMID 19540060
- [Result] Eisbruch A, Harris J, Garden A, et al.: Phase II multi-institutional study of IMRT for oropharyngeal cancer (RTOG 00-22): early results. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-79, S46-7, 2006.
- [Derived] Garden AS, Harris J, Eisbruch A, Chao KSC, Morrison WH, Harari PM, Swanson TA, Jones CU, Yom SS, Spencer SA, Scrimger R, Shenouda G, Shukla M, Lau HY, Mierzwa M, Torres-Saavedra P, Le QT. Final Report of NRG Oncology RTOG 0022: A Phase 1/2 Study of Conformal and Intensity Modulated Radiation for Oropharyngeal Cancer. Int J Radiat Oncol Biol Phys. 2023 Oct 1;117(2):333-340. doi: 10.1016/j.ijrobp.2023.02.057. Epub 2023 Mar 15. No abstract available. PMID 36925074